CLINICAL TRIAL: NCT03420742
Title: A Phase 1 Drug-Drug Interaction Study Between Brigatinib and the CYP3A Substrate Midazolam in Patients With ALK-Positive or ROS1-Positive Solid Tumors
Brief Title: A Phase 1 Drug-Drug Interaction Study Between Brigatinib and the CYP3A Substrate, Midazolam, in Participants With ALK-Positive or ROS1-Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: Brigatinib-1001; U1111-1203-0166 (Other: WHO); 2018-001624-19 (EudraCT Number)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Advanced ALK+ or ROS1+Non-Small-Cell Lung, Neoplasm, Advanced ALK+ or ROS1+Solid Tumors
Keywords: Drug therapy, brigatinib, lung cancer, ALK, ROS1
MeSH Terms: conditions — Carcinoma; Neoplasms; Lung Neoplasms | interventions — Midazolam; brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam 3 mg + Brigatinib 90 mg (Experimental): Midazolam 3 mg, orally, once on Day 1, followed by brigatinib 90 mg, orally, once daily on Days 2 to 8, further followed by brigatinib 180 mg, orally, once daily on Days 9 to 28 in Part A Cycle 1 (28 days treatment cycle). Participants escalating to brigatinib 180 mg once daily will also receive midazolam 3 mg, orally, once on Day 21 of Part A Cycle 1. After completion of Part A, participants will continue into Part B. Participants in Part B will receive brigatinib up to 180 mg (or at the highest tolerated dose in Part A), orally, once daily in a 28 day treatment cycle, up to a maximum of 23 cycles or until progression of disease, unacceptable toxicity, or another discontinuation criterion is met.
  Interventions: Drug: Midazolam; Drug: Brigatinib

INTERVENTIONS:
Drug: Midazolam — Midazolam syrup.
Drug: Brigatinib — Brigatinib tablets.
  Other Names: Alunbrig

SUMMARY:
The purpose of this study is to characterize the effect of repeat-dose administration of brigatinib 180 milligram (mg) once daily (QD) on the single-dose pharmacokinetics (PK) of midazolam.

DETAILED DESCRIPTION:
The study will enroll approximately 20 participants to achieve approximately 15 PK-evaluable participants for assessment. This study will consist of 2 parts: Part A of the study will evaluate the effect of repeat-dose administration of brigatinib on the single-dose PK of midazolam. Part B of the study is exploratory and will allow participants to continue brigatinib until disease progression (PD). All participants will receive study drug via the oral route. Participants will be assigned to: Midazolam 3 mg + Brigatinib 90 mg.

The overall time to participate in this study is 26 months. Participants will have a 28-day PK cycle in Part A and a maximum of 23 cycles in Part B, and a 30-day follow-up period after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic solid tumors who meet 1 of the following 4 criteria:

   * With locally advanced or metastatic ALK-positive NSCLC who have progressed on or are intolerant to treatment with at least 1 other ALK inhibitor.
   * With ALK-positive nonlung solid tumors that are locally advanced or metastatic and for whom no standard, nonexperimental therapy is available.
   * With locally advanced or metastatic ROS1-positive NSCLC who have progressed on crizotinib therapy or are intolerant to crizotinib, or
   * With ROS1-positive nonlung solid tumors that are locally advanced or metastatic and for whom no standard, nonexperimental therapy is available.
2. Eastern cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. Have at least 1 target lesion per response evaluation criteria in solid tumors (RECIST) version 1.1.
4. Have recovered from toxicities related to prior anticancer therapy to National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) version 4.03 Grade less than or equal to (<=) 1.
5. Suitable venous access for study-required blood sampling (that is, including PK and laboratory safety tests).

Exclusion Criteria:

1. Systemic treatment with strong or moderate cytochrome P450 3A (CYP3A) inhibitors or inducers within 14 days before enrollment.
2. Prior therapy with brigatinib.
3. Received prior ALK-inhibitor therapy within 7 days before the first dose of study drug.
4. Treatment with any investigational systemic anticancer agents within 14 days or 5 half-lives, whichever is longer, before the first dose of study drug.
5. Received chemotherapy or radiation therapy within 14 days before the first dose of study drug, except for stereotactic radiosurgery (SRS) or stereotactic body radiation therapy.
6. Received antineoplastic monoclonal antibodies within 30 days before the first dose of study drug.
7. Had major surgery within 30 days before the first dose of study drug. Minor surgical procedures, such as catheter placement or minimally invasive biopsies, are allowed.
8. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Patients with leptomeningeal disease and without cord compression are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- France (2):
  - Hopital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Groupe Hospitalier Bichat-Claude Bernard - Hopital Bichat, Paris, Île-de-France Region
- Italy (6):
  - Centro di Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Santa Maria delle Croci, Ravenna
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands
- Spain (5):
  - Hospital Universitario Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - HM Centro Integral Oncologico Clara Campal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hanley MJ, D'Arcangelo M, Felip E, Garrido P, Zhu J, Ye M, Vranceanu F, Gupta N. A Phase 1 Drug-Drug Interaction Study Between Brigatinib and the CYP3A Substrate Midazolam in Patients With ALK-Positive or ROS1-Positive Solid Tumors. J Clin Pharmacol. 2023 May;63(5):583-592. doi: 10.1002/jcph.2198. Epub 2023 Jan 27. PMID 36579743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the Netherlands, Italy, and Spain from 26 June 2019 to 29 April 2021.
Pre-assignment Details: Participants with anaplastic lymphoma kinase-positive (ALK-positive) or ROS1-positive solid tumors, including non-small-cell lung cancer (NSCLC) were enrolled in this two-part study to receive midazolam with and without repeated doses of brigatinib in Part A, and further continued treatment with brigatinib at their highest tolerated dose (up to 180 milligram [mg]) in Part B. As planned, combined safety data for Parts A and B were collected and reported.
Groups:
- Parts A and B: All Participants: Midazolam 3 mg, oral solution, once on Day 1, followed by brigatinib 90 mg, tablet, orally, once daily on Days 2 through 8, further followed by dose escalation to brigatinib 180 mg, tablet, orally, once daily on Days 9 through 28 in Treatment Cycle 1 (28-day single treatment cycle) in Part A. Participants also received midazolam 3 mg, oral solution, once on Day 21 in Treatment Cycle 1 in Part A. Participants from Part A may have continued into Part B to receive brigatinib 180 mg or their highest tolerated dose received at the end of Part A, tablet, orally once daily in 28-day treatment cycles from Treatment Cycle 2 up to Treatment Cycle 20, or until PD, intolerable toxicity, or another discontinuation criterion was met.
Period: Part A (Cycle 1)
Arm/Group | Parts A and B: All Participants
Started | 24
Completed | 24
Not Completed | 0
Period: Part B (Cycle 2 to Cycle 20)
Arm/Group | Parts A and B: All Participants
Started | 22 (These were the eligible participants from Part A who had the option to continue their treatment in Part B.)
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least 1 dose of any study drug (brigatinib or midazolam).
Arm/Group | Parts A and B: All Participants
Number analyzed (Participants) | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 11
  Netherlands | 2
  Spain | 11
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: Unit: milliliter per minute per 1.73 square meter (mL/min/1.73 m^2).
  mL/min/1.73 m^2 | 97.94 (40.596)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.7 (9.64)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.82 (22.415)

OUTCOME MEASURES:

1. Primary Outcome: Part A, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Midazolam
Description: The statistical analysis was calculated via a mixed-effects analysis of variance (ANOVA) fitting terms for treatment (midazolam with or without brigatinib coadministration).
Time Frame: Cycle 1, Days 1 (Midazolam alone) and 21 (Midazolam + Brigatinib): pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length is 28 days)
Population: PK-evaluable population: participants who received protocol-specified regimen during Part A (including brigatinib 180 mg) without dose reductions/interruptions, did not receive any excluded concomitant medications through completion of PK sampling and had sufficient midazolam concentration-time data to estimate PK parameters by noncompartmental analysis methods. As planned, OM was assessed for Part A only. Overall number of participants analyzed were participants who were evaluable for this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Part A, Cycle 1 Day 1: Midazolam Alone: Midazolam 3 mg, oral solution, once on Day 1 in Treatment Cycle 1 (28-day single treatment cycle) in Part A.
- Part A, Cycle 1 Day 21: Midazolam + Brigatinib: Midazolam 3 mg, oral solution, once along with brigatinib 180 mg, tablet, orally, once on Day 21 in Treatment Cycle 1 (28-day single treatment cycle) in Part A.
Arm/Group | Part A, Cycle 1 Day 1: Midazolam Alone | Part A, Cycle 1 Day 21: Midazolam + Brigatinib
Number analyzed (Participants) | 15 | 14
hour*nanogram per milliliter (h*ng/mL) | 57.2 (30.3) | 42.1 (54.2)
Statistical Analysis 1: Comparison: Part A, Cycle 1 Day 1: Midazolam Alone vs Part A, Cycle 1 Day 21: Midazolam + Brigatinib; Test type: Other; Geometric least squares mean ratio = 0.741, 90% CI 2-sided [0.600 to 0.915] — The ratios of geometric mean were calculated on the basis of the within-participant variance. Participant was treated as a random effect in the model

2. Primary Outcome: Part A, Cmax: Maximum Observed Plasma Concentration for Midazolam
Description: The statistical analysis was calculated via a mixed-effects ANOVA fitting terms for treatment (midazolam with or without brigatinib coadministration).
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK)-evaluable population: participants who received protocol-specified regimen during Part A (including brigatinib 180 mg) without dose reductions/interruptions, did not receive any excluded concomitant medications through completion of PK sampling, and had sufficient midazolam concentration-time data to estimate PK parameters by noncompartmental analysis methods. As planned, this outcome measure (OM) was assessed for Part A only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A, Cycle 1 Day 1: Midazolam Alone | Part A, Cycle 1 Day 21: Midazolam + Brigatinib
Number analyzed (Participants) | 15 | 15
nanogram per milliliter (ng/mL) | 19.7 (42.6) | 16.5 (49.9)
Statistical Analysis 1: Comparison: Part A, Cycle 1 Day 1: Midazolam Alone vs Part A, Cycle 1 Day 21: Midazolam + Brigatinib; Test type: Other; Geometric least squares mean ratio = 0.836, 90% CI 2-sided [0.662 to 1.06] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Part A, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Midazolam
Time Frame: as for outcome 1
Population: PK-evaluable population: participants who received protocol-specified regimen during Part A (including brigatinib 180mg) without dose reductions/interruptions, did not receive any excluded concomitant medications through completion of PK sampling and had sufficient midazolam concentration-time data to estimate PK parameters by noncompartmental analysis methods. As planned, OM was assessed for Part A only.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A, Cycle 1 Day 1: Midazolam Alone | Part A, Cycle 1 Day 21: Midazolam + Brigatinib
Number analyzed (Participants) | 15 | 15
hour | 0.500 [0.220 to 1.93] | 0.500 [0.250 to 1.00]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were adverse events (AEs) that started from the first dose of the study drug up to 30 days after the last dose of the study drug (up to Cycle 20 Day 30 ) (Cycle length =28 days)
Description: Primary objective and endpoint was PK. No secondary objectives/endpoints in study. Part B was exploratory and allowed participants to continue brigatinib therapy to receive potential therapeutic benefits until PD. Since treatment with brigatinib was intended to continue without any modification from Part A into Part B (unless dose modifications were required by toxicity/AE /as indicated by study protocol), therefore it was planned to analyze the combined safety data (Parts A and B).
Arm/Group | Parts A and B: All Participants
All-Cause Mortality (participants affected / at risk) | 8/24
Serious Adverse Events (participants affected / at risk) | 17/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A and B: All Participants (N=24)
Bile duct obstruction (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 1
Confusional state (Psychiatric disorders) | 1
Disease progression (General disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Infection (Infections and infestations) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Parts A and B: All Participants (N=24)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 7
Amylase increased (Investigations) | 5
Anaemia (Blood and lymphatic system disorders) | 7
Aspartate aminotransferase increased (Investigations) | 8
Asthenia (General disorders) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 4
Blood creatine phosphokinase increased (Investigations) | 11
Blood lactate dehydrogenase increased (Investigations) | 2
Chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 9
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 4
Headache (Nervous system disorders) | 3
Hypertension (Vascular disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Lipase increased (Investigations) | 6
Nausea (Gastrointestinal disorders) | 11
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pyrexia (General disorders) | 5
Stomatitis (Gastrointestinal disorders) | 2
Tachycardia (Cardiac disorders) | 2
Urinary tract infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT03420742/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03420742/SAP_001.pdf